CLINICAL TRIAL: NCT02587702
Title: Influence of Improved Formula on Fatty Acids and Mineral Metabolism in Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beingmate Baby & Child Food Co Ltd . (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: RDM2012002
Record Dates: First submitted 2015-10-20; First posted 2015-10-27 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
Keywords: Term Infants
MeSH Terms: interventions — Milk, Human

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Improved Infant Formula Group (Experimental): Containing β-Palmitate Content
  Interventions: Other: β-Palmitate Content
- General Infant Formula Group (Placebo Comparator): Excluding β-Palmitate Content
  Interventions: Other: Placebo
- Human Milk Group (Active Comparator): Containing β-Palmitate Content Naturely in Human Milk
  Interventions: Other: β-Palmitate Content Naturely in Human Milk

INTERVENTIONS:
Other: β-Palmitate Content
  Arms: Improved Infant Formula Group
Other: Placebo
  Arms: General Infant Formula Group
Other: β-Palmitate Content Naturely in Human Milk
  Arms: Human Milk Group

SUMMARY:
The purpose of this study is to determine whether different content of β-palmitate will cause significant differences on Fatty Acids and Mineral Metabolism in Infants

ELIGIBILITY:
Inclusion Criteria:

* Healthy full term infants

Exclusion Criteria:

* experienced congenital or chromosomal disorders
* neonatal morbidities, or metabolic illness

Max Age: 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Content of fatty acids | 3 years
Content of calcium and magnesium | 3 years

SECONDARY OUTCOMES:
Anthropometric measurements | 3 years
  Index of anthropometric measurements contains weight,height and head circumference.
Stool characteristics assessed via stool frequency | 3 years
Stool characteristics assessed via stool consistency | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Children's Medical Center, Shanghai, China